CLINICAL TRIAL: NCT06638970
Title: Clinical Utility and Safety of Human Umbilical Cord Mesenchymal Stem Cell Secretome in Drug Resistant Epilepsy Single Center, Non-randomized, Phase I Clinical Trial
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baermed (Other)
Collaborators: Tarumanagara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001-UTHREC/UNTAR/I/2024
Record Dates: First submitted 2024-10-06; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Epilepsy; Drugs Resistant Epilepsy
Keywords: secretome; stem cells; epilepsy; drug resistant epilepsy; qEEG
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy | interventions — Secretome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Secretome Injection (Experimental): patient will receive 4 times secretome injection every two weeks for two months
  Interventions: Drug: Secretome
- Best Treatment Practice (No Intervention): patient will receive standart therapy for four months

INTERVENTIONS:
Drug: Secretome — 3 ml Injection of secretome for 4 times two weeks apart
  Arms: Secretome Injection

SUMMARY:
The goal of this clinical trial is to learn if Human Umbilical Cord Mesenchymal Stem Cell (HUCMSC) derived secretome injection is safe and effective in patient with epilepsy. The main questions it ams to answer are:

1. How is the relationship between secretome therapy and the reduction in seizure frequency and duration in patients with drug-resistant epilepsy in the adult age group?
2. How does secretome therapy affect EEG and qEEG results in patients with drug-resistant epilepsy in the adult age group?
3. How is the relationship between secretome therapy and the Mini Mental State Examination (MMSE) score in patients with drug-resistant epilepsy in the adult age group?
4. How does secretome therapy affect stress levels as measured by the Perceived Stress Scale (PSS) in patients with drug-resistant epilepsy in the adult age group?
5. How does secretome therapy affect Gait Deviation Index (GDI) scores in patients with drug-resistant epilepsy in the adult age group?
6. How does secretome therapy affect quality of life as measured by the Quality of Life in Epilepsy Inventory (QOLIE-31) in patients with drug-resistant epilepsy in the adult age group?

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 to 60 years.
* Individuals with a clinical diagnosis of epilepsy confirmed by a neurologist based on internationally accepted criteria.
* Individuals with a seizure frequency of at least 6 times in 12 months.
* Individuals who have a history of recurrent seizures that are not controlled with standard antiepileptic treatment of at least 2 types of drugs for at least 12 months.
* Individuals who are in stable general health, without life-threatening acute illnesses or uncontrolled medical conditions.
* Individuals who do not have a history of other neurodegenerative diseases or severe psychiatric disorders that could affect the results of the study.
* Individuals who are not pregnant or breastfeeding.
* Individuals who are willing to provide written consent after receiving complete information about the study.

Exclusion Criteria:

* Individuals with a history of stroke or evidence of stroke on medical examination.
* Individuals who have undergone surgery for the treatment of epilepsy.
* Individuals with a history of allergy or hypersensitivity reactions to the secretome or related components.
* Individuals with active or uncontrolled autoimmune disease.
* Individuals receiving immunosuppressive therapy.
* Individuals with severe hepatic or renal impairment.
* Individuals with significant vascular or blood vessel disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes frequency and duration of the seizures in drugs resistant epilepsy after two months secretome injections | From enrollment to the end of treatment at 2 months, From enrollment to the end of study at 8 months
  Patients achieved a response if there are changes in frequency and duration of the seizures in drugs resistant epilepsy after two months secretome injections.Best outcome when the frequency and duration of the seizures less frequent, worst outcome when the frequency and duration of the seizures get more frequent
Changes in EEG and qEEG (Alpha,Beta, Delta, and Theta wave) results of drugs resistant epilepsy after two months secretome injections | From enrollment to the end of treatment at 2 months, From enrollment to the end of study at 8 months
  Patients achieved a response if there are changes in EEG and qEEG (Alpha,Beta, Delta, and Theta wave) results in drugs resistant epilepsy after two months secretome injections.Best outcome when the EEG and qEEG (Alpha,Beta, Delta, and Theta wave) get a better results, worst outcome when EEG and qEEG (Alpha,Beta, Delta, and Theta wave) get a worse results

SECONDARY OUTCOMES:
Changes in Mini Mental State Examination (MMSE) results of drugs resistant epilepsy after two months secretome injections | From enrollment to the end of treatment at 2 months, From enrollment to the end of study at 8 months
  Patients achieved a response if there are changes in Mini Mental State Examination (MMSE) results in drugs resistant epilepsy after two months secretome injections.Best outcome when the Mini Mental State Examination (MMSE) get a increase results, worst outcome when Mini Mental State Examination (MMSE) get a decrease results
Changes in Perceived Stress Scale (PSS) results of drugs resistant epilepsy after two months secretome injections | From enrollment to the end of treatment at 2 months, From enrollment to the end of study at 8 months
  Patients achieved a response if there are changes in Perceived Stress Scale (PSS) results in drugs resistant epilepsy after two months secretome injections.Best outcome when the Perceived Stress Scale (PSS) get a increase results, worst outcome when Perceived Stress Scale (PSS) get a decrease results
Changes in Gait Deviation Index (GDI) results of drugs resistant epilepsy after two months secretome injections | From enrollment to the end of treatment at 2 months, From enrollment to the end of study at 8 months
  Patients achieved a response if there are changes in Gait Deviation Index (GDI) results in drugs resistant epilepsy after two months secretome injections.Best outcome when the Gait Deviation Index (GDI) get a increase results, worst outcome when Gait Deviation Index (GDI) get a decrease results

OTHER OUTCOMES:
Changes in Quality of The Life in Epilepsy Inventory (QOLIE-31) results of drugs resistant epilepsy after two months secretome injections | From enrollment to the end of treatment at 2 months, From enrollment to the end of study at 8 months
  Patients achieved a response if there are changes in Quality of The Life in Epilepsy Inventory (QOLIE-31) results in drugs resistant epilepsy after two months secretome injections.Best outcome when the Quality of The Life in Epilepsy Inventory (QOLIE-31) get a increase results, worst outcome when Quality of The Life in Epilepsy Inventory (QOLIE-31) get a decrease results

CONTACTS AND LOCATIONS:
Locations (1):
- Main Clinic Prof. Dadang Hawari, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Case Report Form (all collected IPD)
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After publication with no end date

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/24145073/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32577498/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26385090/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/23458467/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34029996/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26302787/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28276062/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7575300/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30426482/
- See also: Related Info — https://medcraveonline.com/JSRT/autologous-bone-marrow-derived-mononuclear-cells-for-the-treatment-of-drug-resistant-epilepsy.html
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29279892/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3348850/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/15950714/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30412924/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/17295717/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/20227351/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/24395517/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/19633196/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31400269/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30140987/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30384669/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30524358/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8661413/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7786246/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27599210/
- See also: Related Info — https://www.researchgate.net/publication/370233760_Quantitative_Electroencephalography_Findings_in_Treatment-resistant_and_Responsive_Patients_with_Idiopathic_Generalized_Tonic-Clonic_Epilepsy
- See also: Related Info — https://www.sciencepublishinggroup.com/article/10.11648/j.ijn.20180201.11
- See also: Related Info — https://www.intechopen.com/chapters/73674
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/21514181/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/24846350/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35206651/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32153072/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35851014/
- See also: Related Info — https://www.researchgate.net/publication/349693823_Hurst_Exponent_and_Tsallis_Entropy_Markers_for_Epileptic_Detection_from_Children
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29588996/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37073101/
- See also: Related Info — https://www.jepilia.org/journal/view.php?number=38
- See also: Related Info — https://paediatricaindonesiana.org/index.php/paediatrica-indonesiana/article/view/2225
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8236431/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37048584/
- See also: Related Info — https://www.swisshealthweb.ch/fileadmin/assets/SANP/2019/sanp.2019.03072/sanp-2019-03072.pdf
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10472368/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31253548/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30974349/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/24286801/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26384579/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32977984/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/19265660/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28316123/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/20525442/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29475054/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/21708072/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/20080419/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/21718708/